CLINICAL TRIAL: NCT00001172
Title: Visual Motor Coordination in Man
Brief Title: Visual Stimulus and Eye Movement
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 800093; 80-EI-0093
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-06

CONDITIONS: Healthy
Keywords: Vision; Eye Movement; Perception; Healthy Volunteer

SUMMARY:
This study is designed to understand how we see visual patterns and how these patterns lead to eye movements.

Normal volunteers participating in this study face a screen on which spots or patterns of light are projected. They are asked to respond to the patterns by voice, eye movements or hand movements. Eye and lid movements are recorded in one of the following ways:

1. Electro-oculogram < small disc electrodes taped to the skin near each eye measure the eye movements as the eyes change position.
2. Infrared detector < an infrared beam is reflected off the eye and picked up by detectors that record the eye movements.
3. Contact lens ring < a smooth plastic ring is placed on the white of the eye surrounding the cornea and eye position is measured using a magnetic coil.

Study sessions last less than four hours.

DETAILED DESCRIPTION:
The purpose of this protocol is to study the physiology of the visuo-motor system in normal humans. This will be accomplished by recording eye movements and other responses (such as reaction time to bar press or verbal responses) to differing stimuli. The stimuli will be primarily visual but may include auditory or tactile stimuli.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal adult volunteers age 18 and over are included.

Only normal volunteers are studied under this protocol. Normal volunteers are recruited from the NIH volunteer office and the NIH web page. Women and minorities are actively recruited.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225
Dates: Start 1980-08-26; Study Completion 2008-08-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Miles FA. The neural processing of 3-D visual information: evidence from eye movements. Eur J Neurosci. 1998 Mar;10(3):811-22. doi: 10.1046/j.1460-9568.1998.00112.x. PMID 9753150
- [Background] Busettini C, Masson GS, Miles FA. Radial optic flow induces vergence eye movements with ultra-short latencies. Nature. 1997 Dec 4;390(6659):512-5. doi: 10.1038/37359. PMID 9394000
- [Background] Masson GS, Busettini C, Miles FA. Vergence eye movements in response to binocular disparity without depth perception. Nature. 1997 Sep 18;389(6648):283-6. doi: 10.1038/38496. PMID 9305842